CLINICAL TRIAL: NCT03731832
Title: Pomalidomide, Ixazomib, and Dexamethasone (PId) With or Without Intensification by Cyclophosphamide (PICd): A Phase II Study in Relapsed or Refractory Multiple Myeloma
Brief Title: Pomalidomide, Ixazomib, and Dexamethasone With or Without Intensification by Cyclophosphamide in Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GWT-TUD GmbH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: DSMM XV
Record Dates: First submitted 2018-10-01; First posted 2018-11-06 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; pomalidomide; Dexamethasone; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: All patients receive PId. Patients showing a biochemical relapse receive PICd afterwards, while patients showing a clinical relapse go off study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PId (Experimental): Treatment of eligible patients with combination of Pomalidomide, Ixazomib, Dexamethasone for all patients until disease progression.
  Interventions: Drug: MLN9708; Drug: Pomalidomide 4 MG Oral Capsule; Drug: Dexamethasone
- PICd (Experimental): Treatment of patients showing an isolated biochemical relapse at disease progression with combination of Pomalidomide, Ixazomib, Dexamethasone plus Cyclophosphamide.
  Interventions: Drug: MLN9708; Drug: Pomalidomide 4 MG Oral Capsule; Drug: Dexamethasone; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: MLN9708 — Study drug will be given as a single, oral dose of 4.0 mg weekly (day 1, 8 and 15) for 3 weeks, followed by 1 week without study drug in a 28-day cycle
  Other Names: Ixazomib 4.0 mg
Drug: Pomalidomide 4 MG Oral Capsule — Study drug will be given as an oral dose of 4.0 mg on day 1 until day 21, followed by 1 week without study drug in a 28-day cycle.
Drug: Dexamethasone — Dexamethasone will be administered as a single, oral dose of 40 mg/day weekly on day 1, 8, 15 and 22 in patients from 18 to 74 years old. For patients ≥ 75 years old dose has to be reduced to 20 mg/day with the same treatment schedule.
Drug: Cyclophosphamide — Cyclophosphamide will be administered once daily as an oral dose of 50 mg on cycle days 1 to 21, followed by one week without drug in a 28-day cycle.
  Arms: PICd

SUMMARY:
The study is designed as a multicenter, non-randomized, Phase II trial with one treatment arm. A total of 82 patients of both genders and older than 18 years with relapsed/refractory multiple myeloma are planned to be included in the study. After the first 6 patients will have finished the first treatment cycle of the induction phase the DMC will assess safety and tolerability of the treatment schedule and decide about the further continuation of the study.

DETAILED DESCRIPTION:
The study is designed as an open-label, non-randomized, multicenter study to investigate the clinical activity of pomalidomide administered once daily in combination with oral ixazomib and dexamethasone (PId) until disease progression according to IMWG criteria.

Patients with clinical relapse (any one of the following: deterioration of renal function, hypercalcemia, newly developing osteolytic lesions and/or soft tissue plasmacytomas) will go off study and receive further treatment according to their treating physician. Patients with isolated biochemical relapse with an increase of serum M-protein of ≥ 25% (absolute increase in serum must be ≥ 5 g/L) and/or urine M-protein (absolute increase in urine must be ≥ 200 mg/24h) or in the difference between involved and uninvolved FLC levels (provided, the absolute increase is > 100 mg/L) without further signs or symptoms will proceed to the intensification phase (PICd).

The intensification phase (PICd) will last until further disease progression. In case of significant haematological and non-haematological toxicities, dose adjustments and/or interruption of the study drugs may be necessary.

Response assessments will be performed every four weeks by evaluation of serum and 24 hour urine specimens. "Progressive disease" (PD) will require a consecutive confirmatory measurement.

ELIGIBILITY:
Inclusion criteria:

* Male or female patients ≥ 18 years of age at the time of signing the informed consent form
* Patients capable to understand the purposes and risks of the study, who are willing and able to participate in the study and from whom written and dated informed consent to participate in the study has been obtained prior to any study related assessments/ procedures being conducted
* Patients with relapsed or refractory, histologically confirmed multiple myeloma
* Patients must have received at least two but not more than four prior anti-myeloma regimens including lenalidomide and bortezomib and have demonstrated disease progression on the last therapy
* Prior treatments must have included both lenalidomide and bortezomib: at least two consecutive cycles of lenalidomide and bortezomib (alone or in combination) and adequate prior alkylator exposure. This is either as part of a stem cell transplant or at least 6 consecutive cycles of an alkylator-based therapy.
* Patients must have failed bortezomib and lenalidomide therapy: progression within 60 days; PR or better with progression within 6 month and/or bortezomib intolerant after ≥ 2 cycles and achieving ≤ MR
* Relapsed from or refractory to at least one regimen (induction, autologous stem cell transplantation (or allogenic stem cell transplantation) and consolidation/maintenance are considered one "regimen")
* Measurable levels of serum and/or urine M-protein: serum M-protein ≥ 5 g/L and/or urine M-protein ≥ 200 mg/24h or serum free light chain (sFLC) concentration of > 100 mg/L of the involved FLC, provided sFLC ratio is abnormal (sFLC K/λ ratio (< 0.26 or > 1.65)
* Life expectancy ≥ 3 months
* ECOG performance status of 0, 1, or 2
* Patients must be able to adhere to the study visit schedule and other protocol requirements
* All women and men must acknowledge to have understood the hazards and necessary precautions associated with the use of pomalidomide and ixazomib
* All subjects must agree in writing to strictly adhere to the Pomalidomide Pregnancy Prevention Plan as given in Appendix C
* Females of childbearing potential (FCBP) must:
* Understand the potential teratogenic risk to the unborn child
* Agree to utilize two reliable forms of contraception simultaneously without interruption for at least 28 days before starting study drug, while participating in the study (including dose interruptions), and for at least 90 days after study treatment discontinuation
* Be capable of complying with effective contraceptive measures
* Be informed and understand the potential consequences of pregnancy and the need to notify her study doctor immediately if there is a risk of pregnancy
* Understand the need to commence the study treatment as soon as study drug is dispensed following a negative pregnancy test
* Understand the need and accept to undergo pregnancy testing based on the frequency outlined in this protocol
* Females must agree to abstain from breastfeeding during study participation and for at least 28 days after study drug discontinuation
* Males must agree to use a latex condom during any sexual contact with FCBP while participating in the study and for 90 days following discontinuation from this study, even if he has undergone a successful vasectomy
* Males must also agree to refrain from donating semen or sperm while on the study drugs and for 90 days after discontinuation from this study treatment
* Subjects must agree to refrain from donating blood while on study therapy and for 28 days after discontinuation from this study treatment
* Subjects must agree not to share medication
* Patients must meet the following clinical laboratory criteria:
* Absolute neutrophil count (ANC) 1 x 109/L
* Platelet count 75 x 109/L for patients in whom < 50% of bone marrow nucleated cells are plasma cells
* Platelet count ≥ 30 x 109/L for patients in whom ≥ 50% of bone marrow nucleated cells are plasma cells. (Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment)
* Total bilirubin 1.5 the upper limit of the normal range (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) 3 ULN
* Calculated creatinine clearance 30 mL/min

Exclusion criteria:

* Concomitant cancer chemo- or radiotherapy (except for local radiation therapy for preexisting lytic lesions)
* Treatment with any investigational product within 60 days prior to first administration of pomalidomide and ixazomib
* Patients eligible for autologous and / or allogeneic stem cell transplantation
* Abnormal/inadequate organ or bone marrow function as defined below (any single parameter to fulfill condition): ANC < 1 x 109/L
* Hemoglobin < 8.0 g/dL (prior RBC transfusion or recombinant human erythropoietin use is permitted)
* Platelet count < 75 x 109/L for patients in whom < 50% of bone marrow nucleated cells are plasma cells
* Platelet count < 30 x 109/L for patients in whom ≥ 50% of bone marrow nucleated cells are plasma cells
* Estimated GFR (MDRD) < 45 ml/min
* AST/ALT > 3 x upper limit of normal (ULN)
* Serum (total) bilirubin > 1.5 x ULN
* Corrected serum calcium > 14 mg/dL (> 3.5 mmol/L); or free ionized calcium > 6.5 mg/dL (> 1.6 mmol/L)
* Serum creatinine > 1.5 x ULN
* Prior pomalidomide based therapy
* Prior ixazomib based therapy
* Baseline peripheral neuropathy > Grade 1 on clinical examination within 14 days before enrollment
* Active HIV, hepatitis B (including patients who are tested Anti-HBc-positive and / or HBsAg-positive) or hepatitis C infection after serologic testing
* Any other concurrent disease or medical conditions that are deemed to interfere with the conduct of the study as judged by the investigator
* Known hypersensitivity to pomalidomide and its analogues in general and/or to ixazomib and its analogues or to any other component of study drugs
* Prior malignancy excluding adequately treated with curative intent basal cell or squamous cell skin cancer, in situ cervical, breast or prostate cancer without any evidence of residual disease or requiring anti-cancer treatment < 2 years prior to initiating study treatment
* Patients with congestive heart failure NYHA Class III and IV, cardiac arrhythmias (except atrioventricular block type I and II, atrial fibrillation/flutter, bundle brunch block) or other signs and symptoms of relevant cardiovascular disease
* Pregnant women, nursing mothers, lactating women, and women of childbearing potential as well as male subjects who are unwilling to adhere to the guidelines of the treatment-specific pregnancy prevention program
* Unwilling or unable to follow protocol requirements
* Systemic treatment with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort within 14 days before randomization in the study
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of the study drugs including difficulty swallowing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Overall Response rate (PId) according to the IMWG criteria. | 1 year throughout study completion
  Overall response rate at PId

SECONDARY OUTCOMES:
Disease control rate | 1 year throughout study completion
  Disease control rate in patients receiving PId (at least SD)
Overall response rate | 1 year throughout study completion
  Overall response rate (PR or better) for patients intensified with PICd
Disease control rate in patients intensified with PICd (at least SD) | 1 year throughout study completion
  Disease control rate in patients intensified with PICd (at least SD)
Progression-free survival (PFS) | 1 year throughout study completion
  Progression-free survival (PFS) for patients receiving PId and for patients receiving PICd
Overall survival (OS) | 1 year throughout study completion
  Overall survival (OS)
Subsequent anti-myeloma regimens (including best response) | 1 year throughout study completion
  Best response during induction by PId

OTHER OUTCOMES:
Molecular cytogenetics by FISH analysis | 1 year throughout study completion
  Evaluation of molecular cytogenetic abnormalities
Safety of the dosing regimens and relationship of AEs | 1 year throughout study completion
  Incidence, severity and relationship of AEs/SAEs of the dosing regimens (safety measures)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Knop, Prof., Principal Investigator — Universitätsklinikum Würzburg / Medizinische Klinik und Poliklinik II
Locations (11):
- Germany (11):
  - Klinikum rechts der Isar der TU München / III. Med. Klinik und Poliklinik, Munich, Bavaria
  - phase drei Hämato-Onkologischer Studienkreis am Klinikum Aschaffenburg, Aschaffenburg
  - Sozialstiftung Bamberg / Klinik am Bruderwald, Zentrum für Innere Medizin, Med. Klinik V, Hämatologie und internistische Onkologie, Bamberg
  - Klinikum der Johann Wolfgang Goethe-Universität Frankfurt am Main, Frankfurt am Main
  - Universitätsklinikum Jena / Klinik für Innere Medizin II, Abteilung für Hämatologie und internistische Onkologie, Jena
  - Universitätsklinikum Magdeburg A.Ö.R / Klinik für Hämatologie und Onkologie, Magdeburg
  - Kliniken Ostalb Stauferklinikum Schwäbisch Gmünd, Mutlangen
  - Universitätsklinikum Münster / Medizinische Klinik A, Münster
  - Studienzentrum Onkologie Ravensburg, Ravensburg
  - Universitätsklinikum Ulm / Klinik für Innere Medizin III, Ulm
  - Universitätsklinikum Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No